CLINICAL TRIAL: NCT02453230
Title: The Effect of Light on the Fetal Biophysical Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Principal Investigator, Heather Said, D.O., University of Nebraska
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 17227
Record Dates: First submitted 2015-01-16; First posted 2015-05-25 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- light on (Active Comparator): BPP done with lights on
  Interventions: Behavioral: Lights on
- light off (No Intervention): Biophysical profile examinations done with the light off

INTERVENTIONS:
Behavioral: Lights on — Determine if ambient room light stimulation changes the amount of time required to perform the fetal biophysical profile.
  Arms: light on

SUMMARY:
Since the 1960's, perinatal mortality in the United States has been declining at a steady rate. This decline has thought to be the result of improved surveillance of normal and abnormal fetal behavior and using that information to determine those babies at risk for stillbirth.

There are many tools available for surveillance. One of these tools, the bio-physical profile (BPP), incorporates a non-stress test (NST) with ultrasound assessment of fetal behavior . This test has been used for about the last 30 years with good safety and efficacy. The ultrasound evaluation includes monitoring fetal breathing, fetal gross and fine movement and amniotic fluid evaluation. NST and BPP have been found to have similar ability to predict fetal well-being, with similar safety and ease of performance. Several studies have observed the effect of sound as well as light on the NST and have found that it can shorten testing time without altering its ability to be interpreted properly or affecting fetal safety. However, similar studies have not been done with the BPP. Light stimulation has been proven to be safe for both the mother and the fetus with no harm having been demonstrated when used with NST.

DETAILED DESCRIPTION:
Since the 1960's, perinatal mortality in the United States has been declining at a steady rate. This decline has thought to be the result of improved surveillance of normal and abnormal fetal behavior and using that information to determine those babies at risk for stillbirth.

There are many tools available for surveillance. One of these tools, the bio-physical profile (BPP), incorporates a non-stress test (NST) with ultrasound assessment of fetal behavior . This test has been used for about the last 30 years with good safety and efficacy. The ultrasound evaluation includes monitoring fetal breathing, fetal gross and fine movement and amniotic fluid evaluation. NST and BPP have been found to have similar ability to predict fetal well-being, with similar safety and ease of performance. Several studies have observed the effect of sound as well as light on the NST and have found that it can shorten testing time without altering its ability to be interpreted properly or affecting fetal safety. However, similar studies have not been done with the BPP. Light stimulation has been proven to be safe for both the mother and the fetus with no harm having been demonstrated when used with NST.

Since the 1960's, perinatal mortality in the United States has been declining at a steady rate. This decline has thought to be the result of improved surveillance as well as neonatal and infant care. However, there is still a large percentage of mortality that is related to antenatal fetal and maternal complications. There has been much research in this area, to help predict which fetuses are more likely to have a poor outcome, and may benefit from intervention, such as early delivery. Several tests have been developed to help monitor fetal behavior and differentiate between fetal well-being and identify those at risk for adverse outcomes. Some of these tests include the contraction-stress test (CST) and the bio-physical profile (BPP), which incorporates the NST with ultrasound assessment of fetal behavior. These tests accurately reflect the acid-base status of the fetus as well as the level of fetal oxygenation.

The biophysical profile was originally developed as a method of assessing fetal health and help determine whether or not a complication of pregnancy was severe enough to warrant delivery. The time length needed to complete a biophysical profile is variable. The test is considered completed if the fetus meets all criteria. The test consists of four ultrasound components, and electronic fetal monitoring component: fetal heart rate reactivity by non-stress test, fetal breathing movements, fetal gross body movements, fetal tone/posture and amniotic fluid evaluation.

These components are scored as a "2" for present and "0" if not present. This makes for a maximum score of 10. Scores of 8 or greater are generally considered reassuring. A score of 6 is considered equivocal and requires further evaluation and follow-up. A score of 4 is concerning and delivery plan should be initiated soon. A score of 2 or 0 should means the fetus should be delivered immediately.

Fetal heart rate reactivity is assessed with a fetal non-stress test using a external electronic fetal monitor. The mother has an external tocodynomometer and a small doppler device placed over the area of the fetal chest placed on her abdomen. The test is considered "reactive" when there are two defined accelerations of the fetal heart rate above the baseline rate during the 20 to 30 minute testing period. The size of the acceleration required depends on the gestational age of the fetus. Testing time can be extended up to 60 minutes to obtain reactivity if the fetus happens to be in a passive sleep state during the test.

Fetal breathing movements have been seen by ultrasound beginning in the early second trimester. The consist of intermittent "practice" breathing by the fetus where the diaphragm can be seen moving similarly to adults. These movements last greater than 30 seconds but are not continuous. This is the first finding to be lost when fetal hypoxemia is present.

Body or limb movements are generally decreased in fetuses that are hypoxic. This corresponds to decreased activity level for metabolic conservation in those fetuses that are compromised. Three or more discrete movements are required for this to be considered present.

Fetal tone and posture are demonstration of active extension with rapid return to flexion of fetal limbs and brisk repositioning or trunk rotation. Opening and closing of hand or mouth, kicking, and so on. One example must be observed for this to be considered present during the exam.

Amniotic fluid evaluation is considered present when at least one pocket of fluid is seen on ultrasound measuring greater than 2 centimeters without umbilical cord present.

Response of fetuses to light stimulation has been known since 1975 when Polishuk reporting fetal movement after 26 weeks gestation in fetuses stimulated by light. In 1980, Peleg and Goldman performed amnioscopy and noted an acceleration in the fetal heart rate in 80% of patients after being exposed to the light of the amnioscope. Caridi et al. noted that fetuses stimulated with halogen light took less time to become reactive on a non-stress test than fetuses that were not stimulated. No study has noted an adverse maternal or fetal event from use of light stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Mothers age 14-60 years old with singleton pregnancies at 20 0/7th weeks to 42 6/7th weeks gestational age
* Biophysical testing has been ordered for any indication other than higher order multiple gestations.

Exclusion Criteria:

* Patient declines to participate.
* Multiple gestations (twins or more)

Ages: 14 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Amount of time needed to complete the biophysical profile | Patients to be followed from initiation of biophysical profiles until delivery an expected average of 8 weeks)
  Measure if ambient room light stimulation changes the amount of time required to perform the fetal biophysical profile

CONTACTS AND LOCATIONS:
Overall Officials: Heather Said, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No